CLINICAL TRIAL: NCT03274570
Title: Factors Affecting Hand Dysfunction in Patient With Rheumatoid Arthritis and Its Correlation With Quality of Life
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Essraa Mohammed, Principal Investigator, Assiut University
Other Study IDs: Hand function in RA
Record Dates: First submitted 2017-08-27; First posted 2017-09-07 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — CBC;ESR,liver function test and kidney function test
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aims of the research are:

* To predict factors affecting hand dysfunction in patient with rheumatoid arthritis
* To study the effect of hand dysfunction on quality of life in patient with rheumatoid arthritis

DETAILED DESCRIPTION:
Rheumatoid Arthritis (RA) is the most common chronic autoimmune systemic inflammatory arthritis, associated with considerable impairments of Quality of life .

Hand is the principle means by which an individual interacts with people and objects in the external environment .Many factors affect hand function in addition to arthritis ,. Many RA patients suffer from an increased loss of muscle mass with a significant impact on these patients' quality of life , and also Distal sensory, mixed sensorimotor, mononeuritis multiplex and entrapment neuropathy are the most commonly reported types of neuropathy in RA .So assessment of factors causing hand dysfunction can provide us a quick and early insight on the debilitating effects of RA on functioning and disability.Thus Early intervention can then be initiated which will help limit joint damage and thereby improve functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients who fulfilled the American College of Rheumatology (ACR) (2010) criteria for RA, attending the Rheumatology and Rehabilitation outpatient clinic and in-patient department, Faculty of Medicine, Assuit University Hospitals.

Exclusion Criteria:

* Patients with other rheumatic diseases.
* Patients less than 18 years old.
* Patients with co-morbidities influencing disease activity and hand function (e.g., end- stage liver or renal disease, serious infections, or severe cardiac, respiratory, gastrointestinal disease) .
* Patient with any recent history of hand trauma, or surgery.
* Patient with neurological involvement as , peripheral neuropathy and radiculopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient attending the Rheumatology and Rehabilitation outpatient clinic and in-patient department, Faculty of Medicine, Assuit University Hospitals during the period from September 2017 until September 2018
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-10-30 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
quality of life | one year
  Health assessment questionnaire disability index (HAQ)

SECONDARY OUTCOMES:
hand function | one year
  measured by musculoskeletal ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Safaa A Mahran, professor, Study Director — Assiut University; Essam Abda, professor, Study Director — Assiut University